CLINICAL TRIAL: NCT04937530
Title: A Randomized, Double-blind, Controlled, Phase 2 Study to Assess Efficacy, Long Term Safety and Tolerability of RT001 in Subjects With Progressive Supranuclear Palsy
Brief Title: RT001 in Patients With Progressive Supranuclear Palsy (PSP) PROGRESSIVE SUPRANUCLEAR PALSY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT001-013
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — RT001; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RT001 (Experimental): RT001 960 mg capsule. 3 capsules TID for 4 weeks, followed by 3 capsules BID for the remaining 44 weeks.
  Interventions: Drug: RT001
- Placebo (Placebo Comparator): Inactive comparator capsule 960 mg (safflower oil). 3 capsules TID for 4 weeks, followed by 3 capsules BID for the remaining 44 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RT001 — RT001 8.64 g/d (3 capsules TID) for 1 month followed by 5.76 g/d (3 capsules BID) for an additional 11 months
  Other Names: di-deuterated linoleic acid ester
  Arms: RT001
Drug: Placebo — Placebo Comparator: Placebo Inactive comparator capsule 960 mg/capsule: 3 capsules TID for 4 weeks, followed by 3 capsules BID for the remaining 44 weeks.
  Other Names: safflower oil
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled trial of RT001 in patients with PSP.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled trial of RT001 in patients with PSP to assess the efficacy, safety and tolerability of RT001. Subjects will be randomized to RT001 or placebo and will receive study drug for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form prior to entry into the study
2. Male or female subject with age 40 years to 80 years at the time of signed consent
3. Meets the MDS-PSP study group criteria for possible or probable progressive supranuclear palsy with Richardson syndrome (postural instability and falls with vertical ocular motor dysfunction)
4. Presence of PSP symptoms for less than 4 years
5. Score of <40 on the PSPRS-28
6. Ambulatory patients (with or without assistive device - no handheld help) and capable of performing study assessments/evaluations
7. Subject has an identified, reliable, study partner (e.g., caregiver, family member, social worker, or friend) who can assist in assuring that the subject is able to travel to the required visits.
8. Willing to provide the necessary blood samples

Exclusion Criteria:

1. Received treatment with other experimental therapies within the last 30 days prior to the first dose. The last dose of the prior experimental agent must have occurred more than 5 half-lives prior to enrollment in the current trial.
2. Previously received treatment with RT001
3. Refusal to discontinue fish oils or other oil-based supplements for the duration of the study (Screening/Baseline till last study procedure completed)
4. Mini mental state examination (MMSE) score less than 20 at screening
5. Subject resides at a skilled nursing or dementia care facility, or admission to such a facility is planned during the study period
6. Evidence of any clinically significant neurological disorder other than PSP in particular CBS
7. Evidence of a clear and robust benefit from levodopa at the time of screening. Participants are permitted to take levodopa and other Parkinson's medications if the dose had been stable for 60 days prior to screening
8. The subject has a history of or currently has schizophrenia, schizoaffective disorder or bipolar disorder according to DSM-V or ICD-10 criteria
9. Subject has had a significant illness or infection requiring medical intervention in the past 30 days
10. Subject has evidence of any disease or condition (based on either history, physical or laboratory values) that might interfere with the conduct of the study
11. Is currently receiving active deep brain stimulation (DBS) that cannot be turned off
12. Any condition with a life expectancy of less than 2 years
13. Female who is breastfeeding or has a positive pregnancy test
14. Male participant or female participant of childbearing potential, who is sexually active and unwilling/unable to use a highly effective birth control method throughout the study
15. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to return for visits as scheduled
16. History, within the last 2 years, of alcohol abuse or physical opioid dependence

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the PSPRS-28 at 48 weeks for the RT001 treated group vs placebo-treated group | 48 weeks
  The PSPRS-28 is a clinician-rated instrument to assess disability and severity of PSP. The PSPRS-28 evaluates 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lorenzl, MD, PhD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Agaharied Teaching Hospital, University of Munich, Munich, MD, Germany

IPD SHARING:
Plan to Share IPD: No